CLINICAL TRIAL: NCT02911636
Title: 5 Fractions of Pelvic SABR With Intra Prostatic SABR
Acronym: 5STAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Andrew Loblaw (Other)
Responsible Party: Sponsor-Investigator, Andrew Loblaw, Principal investigator, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 360-2016
Record Dates: First submitted 2016-09-14; First posted 2016-09-22 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Pelvic SABR with intra-prostatic SABR
  Interventions: Radiation: Pelvic SABR with intra-prostatic SABR

INTERVENTIONS:
Radiation: Pelvic SABR with intra-prostatic SABR — described elsewhere

SUMMARY:
Stereotactic Ablative Radiation(SABR) 35 Gy in 5 fractions, once weekly to prostate with simultaneous intraprostatic boost to the MR detected nodule up to 50Gy + 25 Gy in 5 fractions, once weekly simultaneously to seminal vesicles (SV's) and pelvic lymph nodes + 6-18 months of ADT

DETAILED DESCRIPTION:
SABR 25Gy / 5 fractions to pelvis; 35Gy / 5 fractions to prostate; up to 50Gy / 5 fractions to MR nodule

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma (centrally reviewed)
* High- tier intermediate risk defined as:

PSA 10-20ng/ml AND (T2b-2c OR Gleason 7 )

• High-risk prostate cancer, defined as at least one of: T3, OR Gleason 8-10, OR PSA > 20 ng/mL

* Willing to give informed consent to participate in this clinical trial
* Able and willing to complete Expanded Prostate Index Composite (EPIC) questionnaire

Exclusion Criteria:

* Prior pelvic radiotherapy
* Contra-indication to radical prostate radiotherapy e.g. connective tissue disease or inflammatory bowel disease
* Contraindication to prostate MRI
* Anticoagulation medication (if unsafe to discontinue for gold seed insertion)
* Diagnosis of bleeding diathesis
* Large prostate with significant arch interference on TRUS after 3 months of neoadjuvant ADT.
* Previous TURP
* Poor baseline urinary function defined as International Prostate Symptom Score (IPSS) >20
* Significant medical co-morbidity rendering patient unsuitable for general anesthetic
* No evidence of castrate resistance (defined as PSA < 3 ng/ml while testosterone is < 0.7nmol/l. Patients could have been on combined androgen blockade but are excluded if this was started due to PSA progression.
* Definitive extrapelvic nodal or distant metastatic disease on staging investigations.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
To document the number of patients with grade 3 or higher acute urinary and/or bowel toxicity using the Common Terminology Criteria for Adverse Events (CTCAE v4.0) criteria | 3 months after accrual target is reached

IPD SHARING:
Plan to Share IPD: No